CLINICAL TRIAL: NCT05646212
Title: Integrating Treatment for Mental Disorders in Methadone Clinics in Ukraine
Acronym: MEDIUM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ukrainian Institute on Public Health Policy (Other)
Collaborators: Yale University (Other); Alliance for the Public's Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA045384 (NIH)
Record Dates: First submitted 2022-04-08; First posted 2022-12-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Depression; Opioid Use Disorder
Keywords: depression; opioid use disorder; opioid agonist treatment; Ukraine
MeSH Terms: conditions — Depression; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Standard of care (with SSRI medications provided for free).
- SOC+ECHO (Experimental): Standard of care (with SSRI medications provided for free), plus Project ECHO facilitation (an evidence-based tele-education intervention) for physicians
  Interventions: Other: Project ECHO
- SOC+ECHO+P4P (Experimental): Standard of care (with SSRI medications provided for free), plus Project ECHO facilitation (an evidence-based tele-education intervention) for physicians, plus Payment for Performance intervention
  Interventions: Other: Project ECHO; Other: Payment for Performance

INTERVENTIONS:
Other: Project ECHO — Project Extension for Community Healthcare Outcomes® (ECHO): This EBP, tested originally to facilitate HCV care into non-specialty settings, is based on established educational theories of social learning & behavior change in where non-specialists collaborate with specialists, resulting in an innovative healthcare delivery model that results in equivalent quality care for patients in non-specialty settings.
  Arms: SOC+ECHO; SOC+ECHO+P4P
Other: Payment for Performance — P4P in healthcare, endorsed by 3 IOM reports, gives financial incentives to clinicians for adhering to clinical guidelines and achieving better health outcomes. One 2007 IOM report recommended "physician incentives so that profitability and improved healthcare delivery is aligned with patient safety goals and strengthen the business case for healthcare quality and safety."
  Arms: SOC+ECHO+P4P

SUMMARY:
The MEDIUM study (U01DA045384) is a cluster-randomized trial based in Ukraine. The main goal of the study is to test the implementation strategies for mental health treatment services in OAT clinics.

The study enrolled 12 OAT clinics from 12 geographically and epidemiologically diverse regions and randomized them 1:1:1 to three implementation arms: standard of care (SoC), ECHO facilitation, and ECHO plus pay-for-performance (P4P) incentives. Project ECHO, is an evidence-based telehealth intervention, connecting clinicians with national experts for short thematic didactic sessions and case discussions. All sites are provided with a modified Screening, Brief Intervention and Referral to Treatment (mSBIRT) intervention manual for mental disorders and regular supply of two selective serotonin reuptake inhibitors (SSRI) medications. All current and new patients at participating sites (N~2000 at study start) are automatically eligible for SSRI prescription. The main outcomes of the study are the elements of mental health continuum of care (screening, diagnosis, treatment and retention). These outcomes are assessed in the entire patient population using de-personalized data extracted from the electronic medical record system. A sub-sample of patients (N=1,350) was recruited into a cohort and consented to assess prevalence and severity of mental disorders, various factors related to the uptake of and retention in mental health treatment (addiction severity, other substance use, co-morbidities), as well as other important covariates. These assessments are done at baseline, 6, 12, 18 and 24 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving OAT at participating sites

Exclusion Criteria:

* Not willing to participate
* Unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients screened for depression by clinical staff using Patient Health Questionnaire-2 (PHQ-2) | 30 months (August 2019 - February 2022)
  Site-level indicator
Proportion of patients assessed by physician using Montgomery-Asberg Depression Rating Scale (MADRS) and motivated for treatment | 30 months (August 2019 - February 2022)
  Site-level indicator
Proportion of patients initiated on Selective serotonin reuptake inhibitors (SSRIs) | 30 months (August 2019 - February 2022)
  Site-level indicator
Proportion of patients retained on Selective serotonin reuptake inhibitors (SSRIs) | 30 months (August 2019 - February 2022)
  Site-level indicator

SECONDARY OUTCOMES:
Number of participants who continue opioid agonist treatment at the assessment time point | 3, 6, 12, 18 and 24 months after enrollment for each patient
  Retention on opioid agonist treatment
Psychiatric Quality of Life (SF-12 mental component score) changes over time | 3, 6, 12, 18 and 24 months after enrollment for each patient
  Change in the mental component score of the Short-Form Health Survey version 2 (SF-12v2) scale (0-100, higher means better health).

CONTACTS AND LOCATIONS:
Overall Officials: Sergiy Dvoryak, MD, PhD, Principal Investigator — Ukrainian Institute on Public Health Policy
Locations (9):
- Ukraine (9):
  - Kryvyi Rig psycho-neurological dispensary, Kryvyi Rih, Dnipropetrovsk Oblast
  - Dnipropetrovsk narcological dispensary, Pavlohrad, Dnipropetrovsk Oblast
  - Kropyvnitsky regional narcological dispensary, Kropyvnytskyi, Kirovohrad Oblast
  - Mykolaiv regional narcological dispensary, Mykolayiv, Mykolaiv Oblast
  - Ternopil regional narcological dispensary, Ternopil, Ternopil Oblast
  - Ivano-Frankivsk regional narcological dispensary, Ivano-Frankivsk
  - Kyiv city narcological clinic 'Sociotherapia', Kyiv
  - Mykolaiv City Hospital #5, Mykolayiv
  - Vinnitsia regional narcological dispensary 'Sociotherapia', Vinnytsia

IPD SHARING:
Plan to Share IPD: Undecided